CLINICAL TRIAL: NCT00707460
Title: Objective 3: Pilot Dietary Trial; The Sandy Lake Health & Diabetes Project (SLHDP): Understanding and Addressing Metabolic Syndrome, Diabetes and Associated Complications in Aboriginal Canadians
Brief Title: The Effect of a Traditional Dietary Intervention on Diabetes Mellitus and Cardiovascular Disease Risk Factors in a First Nation Community: A Pilot Study
Acronym: SLHDP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Anthony Hanley, PhD, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22419; MOP44076
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; Obesity
Keywords: Diabetes; Cardiovascular; Obesity; First.Nation; Aboriginal (Health); Dietary; Intervention; Nutrition; Traditional (Diet); Sandy Lake (Health & Diabetes Project); (High) protein; (High) fibre (er); (Low) carbohydrate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Diabetes Mellitus | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Please, see design section for details.
  Interventions: Behavioral: Dietary Intervention (Macronutrient composition)
- 2 (Experimental): Traditional Diet
  Please, see design section for details.
  Interventions: Behavioral: Dietary Intervention (Macronutrient composition)
- 3 (Experimental): Healthy Store-bought Diet
  Please, see design section for details.
  Interventions: Behavioral: Dietary Intervention (Macronutrient composition)

INTERVENTIONS:
Behavioral: Dietary Intervention (Macronutrient composition) — The Traditional Diet and Healthy Store-Bought arms differ from the control group and one another by their macronutrient composition. Please, see design section for more detail on this item.
  All groups are exposed to nutrition education on serving size and portion size.
  Other Names: high protein diet = traditional diet; high fiber diet = healthy store-bought diet; high carbohydrate diet = healthy store-bought diet

SUMMARY:
The purpose of this study is to evaluate whether or not a traditional First Nations diet (high protein) and/or a dietary intervention based upon current Canadian dietary recommendations (high carbohydrate/high fiber) effects risk factors for type 2 diabetes mellitus and/or cardiovascular disease in a remote fly in First Nations community (Sandy Lake First Nation).

This pilot has been developed in conjunction with Sandy Lake First Nation to answer the research question: Will a traditional diet or a diet based upon current Canadian dietary recommendations result in decreasing risk for type 2 diabetes in Sandy Lake?

DETAILED DESCRIPTION:
Eligible participants will be randomized to one of 3 groups. Potential participants will have an oral glucose tolerance test (OGTT) during the screening visit to evaluate if they are eligible for the study. Those who meet the inclusion criteria will be stratified according to diagnoses (normal glucose tolerance or impaired glucose tolerance) and randomized to one of three diet groups for a 6 month period.

The following is a description of the 3 study arms/diets:

Group 1: The (Food choice) Control Group

Group 2 (The "Traditional Food" [TD] Group) will receive instruction to follow a diet that reflects the traditional nutrient intake pattern of this population. Briefly, participants will be encouraged to consume, wild meats (i.e. moose, duck, rabbit, and beaver), fish, local berries and other foods obtained from the land ("bush foods"). When these foods are not available, acceptable store bought substitutes will be encouraged (i.e. low fat beef & pork, skinless chicken, canned/frozen fish, store bought fruit and frozen berries). Traditional preparation methods will also be encouraged (i.e. boiling, smoking, and BBQing), and non-traditional foods (i.e. high saturated fat, high carbohydrate, processed foods, high sodium foods, "junk foods", convenience foods or foods including trans fats) and preparation methods (i.e. frying) will be strongly discouraged. The diet has been developed by a Registered Dietitian (RD) with the feedback of Sandy Lake First Nation community members, Dr. Anthony Hanley and with the assistance of tools and documents obtained from Health Canada's website.

Group 3 (The "Healthy Store-bought Food" [HSF] Group) will receive instruction to follow a diet that reflects the results of nutritional epidemiological research on diabetes prevention in this and other populations. Participants will be encouraged to consume a diet comprised of foods as per the Canadian Food Guide to Healthy Eating, Health Canada. It is estimated that HSF group participants will have a macronutrient profile that reflects current "Acceptable Macronutrient Distribution Range (AMDR)", as per the Institute of Medicine (2005) and Health Canada (2007) if they adhere to the education provided. Recommendations will promote a high fibre, low trans- and saturated fat diet including whole grains, fruit and vegetables, mono- and poly-unsaturated fat sources, lean meat and poultry and a low fat dairy profile. "Junk food" (i.e. soda pop, chips, and chocolate bars) will not be forbidden, however will be regarded as a "choose less often" food. Convenience/Ready-Made foods will be allowed, however, healthier choices will be highlighted during the education sessions.

All three groups will be provided with education on serving size and portion control to promote compliance and to ensure that all groups are obtaining useful nutritional information by participating in the study. A major component of the SLHDP is to promote capacity building and long term healthy lifestyle in the community. Portion control will be treated as a controlled variable and will promote identical caloric intake between and within groups.

Nutrition Education and Lifestyle Data Collection:

Community support staff will be trained by the Research Coordinator/ Registered Dietitian (RD) to conduct baseline and follow-up sessions when the RD is not stationed in Sandy Lake. The Research Coordinator/ RD will be available 9am-5pm (week days)for nutrition consult and information support. During follow-up sessions data will be collected (see outcome measures) and data collection tools, food provisions and education will be provided.

Metabolic/Anthropometric Data Collection:

A Community (member) Registered Practical Nurse will be responsible for the metabolic and anthropometric data collection (see outcome measures). This RPN has held this role since the beginning of the SLHDP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Sandy Lake First Nation permanent resident, with total travel outside of the community less than one month per year.
* Aboriginal Ethnicity
* BMI = 23-40 kg/m2
* According to Prochaska and DiClemente's transtheoretical model, also referred to as the Stages of Change Theory, potential participants must be at least at the contemplation stage.
* Willing and able to follow the study protocol

Exclusion Criteria:

* DM detected by OGTT
* Pregnancy, lactation or intention to become pregnant within six months from recruitment
* Any pre-existing condition compromising macronutrient metabolism, quality of life or ability to participate according to protocol. Individuals with the following conditions will be excluded automatically: heart disease, cerebrovascular disease, diagnosed HIV/AIDS, cancer, emphysema, liver or kidney disease
* Insurmountable language barriers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pilot Study: no formal primary outcome measure. There is no noted safety issue for this study; although adverse/side effects and/or symptoms will be closely monitored by the RPN and community research staff. | 6 months

SECONDARY OUTCOMES:
Indicators of glycemic control: fasting blood glucose, insulin resistance, fasting serum insulin, liver function tests, urine creatinine, sodium and other urinary nutritional indicators (from the same urine sample) and full lipid profile. | 6 months
Blood pressure (BP) and heart rate | 6 months
Non-traditional CVD risk factors: serum C-reactive protein (CRP) and adiponectin. | 6 months
Anthropometric measurements: change in body mass (kg)/BMI over the study period, change in percent body fat and percent lean body mass (bio-electrical impedance analysis [BIA]), and waist and hip circumference. | 6 months
Compliance of the sample using three day diet records and appointment attendance. Participants' barriers to compliance will be assessed via the questionnaire(s), diet records and study chart notes. | 6 months
Future dietary intervention feasibility will be assessed by 24-hour recalls/ diet records, appointment attendance, participant and community staff feedback, and questionnaire completion. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, DM, PhD, Study Director — University of Toronto
Locations (1):
- Sandy Lake Health & Diabetes Project Research Office, Sandy Lake, Ontario, Canada